CLINICAL TRIAL: NCT03040323
Title: Prospective Analysis of Value of Contrast-enhanced Sonography During Biopsies of Focal Liver Masses
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient patient recruitment. Data lost following departure of key personnel
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jordan K. Swensson, Assistant Professor Clinical Radiology, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1609504711
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-07

CONDITIONS: Liver Biopsy
MeSH Terms: interventions — Powders; Injections

STUDY DESIGN:
Intervention Model Description: Two interventional arms, selected by day of month; 1) biopsy with Lumason, 2) biopsy with placebos
Who Masked: Participant
Masking Description: Patients will not be informed of diagnostic arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- biopsy with Lumason (Experimental): liver biopsy performed with prior contrast enhancement with Lumason 60.7Mg Powder for Injection (experimental method)
  Interventions: Drug: Lumason 60.7Mg Powder for Injection
- biopsy with placebos (Placebo Comparator): liver biopsy performed without prior contrast enhancement (standard method)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Lumason 60.7Mg Powder for Injection — Lumason 60.7Mg Powder for Injection injected prior to ultrasound-guided biopsy
  Other Names: Lumason
  Arms: biopsy with Lumason
Drug: Placebos — Placebos injected prior to ultrasound-guided biopsy
  Arms: biopsy with placebos

SUMMARY:
The investigators plan to compare complication and success rates between two methods of ultrasound guidance for biopsy of liver lesions, contrast-enhanced and the current protocol without contrast.

DETAILED DESCRIPTION:
As a major oncology and hepatology center, the investigators perform about 3-5 guided biopsies for liver tumors weekly. Ultrasound is the preferred modality for imaging biopsies due to its ability to visualize and position the biopsy needle in real time with high accuracy and safety, is nonionizing, and is quicker compared to other techniques, especially CT-guided biopsies. The failure rate of ultrasound guided liver biopsies (including cases where biopsy was declined to be performed due to lack of lesion visibility) is about 10%. By comparison, in the investigators' practice genotyping of metastatic tumors, with multiple core biopsies, is often requested for entry into oncology trials, and failure of tumor genotyping after biopsy is estimated to be about 30%.

Recently, the first ultrasound contrast agent was FDA-approved for characterization of liver lesions [sulfur hexafluoride lipid-type A microspheres (Lumason, Bracco Diagnostics, Monroe Township, NJ)]. The microbubble agent is deemed safe, including in cardiac failure patients and those with chronic airway obstruction. Injecting microbubbles may allow better visualization of lesions and adjacent vasculature by enhancing the microvasculature and adjacent vessels and potentially reduce incidence of failed biopsy or bleeding complications. In addition, determination of necrotic regions in a lesion may allow better direction of biopsy.

Yet there is limited literature on the use of ultrasound contrast agents for improving targeted liver biopsies. The investigators intend to prospectively assess the non-diagnostic biopsy and complication rates in a group of patients who undergo contrast-enhanced ultrasonography (CEUS) using microbubbles at the time of biopsy. The investigators will then compare the results from this group with the failure and complication rate from a control group of patients undergoing the standard US-guided biopsy procedure. Over 12 months the investigators expect to perform approximately 200 biopsies. Power analysis suggests that 125 patients in both contrast-enhanced sonography and control groups, each, are required. The investigators should be able to enroll sufficient patients in 18 months

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Age 18 years or greater
3. Scheduled to undergo liver biopsy with ultrasound guidance at a performance site

Exclusion Criteria:

1. Liver biopsy is not intended to obtain tissue from a specific lesion
2. Known or suspected cardiac shunt
3. History of hypersensitivity to any active or inactive ingredients in Lumason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kumar Sandrasegaran, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Insufficient patient recruitment and following internal IRB audit study was abandoned/terminated. The PI has left the institution and no information is available regarding how many participants Started and Completed the study in each arm
Groups:
- Biopsy With Lumason: Lumason 60.7Mg Powder for Injection injected prior to ultrasound-guided biopsy
- Biopsy With Placebos: Placebos injected prior to ultrasound-guided biopsy.
Period: Overall Study
Arm/Group | Biopsy With Lumason | Biopsy With Placebos
Started | 0 (No information available regarding how many participants Started and Completed the study in each arm) | 0 (No information available regarding how many participants Started and Completed the study in each arm)
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Insufficient patient recruitment and following internal IRB audit study was abandoned/terminated. The PI has left the institution and it is not clear if Baseline data were collected. No Baseline data are available
Groups:
- Total: Total of all reporting groups
Arm/Group | Biopsy With Lumason | Biopsy With Placebos | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]
Insufficient patient recruitment and data was lost following departure of key study personnel

OUTCOME MEASURES:

1. Primary Outcome: Complication Rate
Description: Complication will be defined as 1) bleeding seen on post-biopsy CT or US, 2) drop in hemoglobin of more than 1.5 g/dL within one week after biopsy, or 3) need for hepatic artery embolization.
Time Frame: 30 days
Population: Insufficient patient recruitment and following internal IRB audit study was abandoned/terminated. No data were collected for Outcome Measures
Groups:
- Biopsy With Lumason: Lumason 60.7Mg Powder for Injection injected prior to ultrasound-guided biopsy;
Arm/Group | Biopsy With Lumason | Biopsy With Placebos
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Success Rate
Description: Biopsy sample being sufficient for histological diagnosis and/or complete genotyping.
Time Frame: 30 days
Population: as for outcome 1
Arm/Group | Biopsy With Lumason | Biopsy With Placebos
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Insufficient patient recruitment and following internal IRB audit study was abandoned.
Description: Insufficient patient recruitment and following internal IRB audit study was abandoned/terminated. The PI has left the institution and no information is available regarding Adverse Events
Arm/Group | Biopsy With Lumason | Biopsy With Placebos
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Insufficient patient recruitment and data was lost following departure of key study personnel

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT03040323/Prot_000.pdf